CLINICAL TRIAL: NCT06781580
Title: The Effectiveness of an Ergonomic Protocol in Reducing Ergonomic Risk and Improving Performance for Competitive E-Sport Athletes
Brief Title: Ergonomic Protocol for Competitive E-Sport Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Donnamarie Krause, Principal Investigator, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNLV-2024-426
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: No Disease or Condition is Being Studied
Keywords: Ergonomics; Esports athletes; Gamers; Gaming; Ergonomic protocol; Musculoskeletal disorders; Ergonomic risk; Performance; Repetitive strain injuries; Accuracy; Aim; Postural rehabilitation; Esports
MeSH Terms: conditions — Musculoskeletal Diseases; Cumulative Trauma Disorders; Episodic Ataxia, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ergonomic Protocol for Esports Athletes (Experimental): This arm of the study involves the implementation of a six-week ergonomic protocol specifically designed for esports athletes who primarily use a PC setup (mouse and keyboard). The intervention includes an educational component on proper posture, warm-ups, and cool-down exercises, as well as a postural rehabilitation program to reduce the risk of repetitive strain injuries and improve gaming performance. Participants will attend four in-person sessions for assessments and training, with ergonomic risk and gaming performance evaluated at baseline, mid-point, and post-intervention. A focus group and long-term follow-up questionnaire will also be included to gather feedback and assess adherence to the protocol.
  Interventions: Other: Esports Ergonomic Protocol

INTERVENTIONS:
Other: Esports Ergonomic Protocol — The Esports Ergonomic Protocol is a six-week intervention designed to reduce the risk of repetitive strain injuries and enhance gaming performance for esports athletes. It includes an educational session on ergonomics, focusing on proper posture, body mechanics, and workstation setup. The protocol also incorporates warm-up and cool-down exercises to prevent strain and improve flexibility, as well as a postural rehabilitation program targeting the upper extremities and core muscles.
  Participants will attend four in-person sessions at specified intervals for ergonomic risk assessments (using REBA) and gaming performance evaluations (using Kovaaks). The intervention also features online resources, including exercise tutorials and ergonomic tips, to support adherence and long-term implementation. Feedback will be collected through post-intervention surveys and an optional focus group to refine the protocol for future use in the esports community.
  Other Names: Gaming Ergonomics Intervention; Ergonomic Training for Esports Athletes

SUMMARY:
The goal of this clinical trial is to learn if this ergonomic protocol can improve performance and reduce ergonomic risk in esports athletes. It will also learn about the insight of esports athletes and their experience in implementing this new protocol. The main questions it aims to answer are:

Does this ergonomic protocol improve performance? Does this ergonomic protocol reduce ergonomic risk?

Researchers will assign the protocol to esports athletes who meet inclusion criteria and express interest in participating in the study. A pre-post design will be conducted to note any differences.

Participants will:

* Participate in a 6-week study with 4 in-person visits
* Volunteers will be requested to participate in a focus group during Week 6.
* Implement the strengthening protocol 3x a week and a warm up/cool down protocol before and after each gaming session.
* Attend one educational session about gaming ergonomics during Week 1
* Complete the Rapid Entire Body Assessment, Kovaaks Asessment, and a Questionnaire during Week Zero, Week 3, and Week 6.

DETAILED DESCRIPTION:
1. Recruitment will occur via snowballing, word-of-mouth, flyers, emails, and social media posts
2. Potential participants will complete a general Demographic questionnaire via Qualtrics as part of the inclusion criteria, collecting information such as age, race, type of gaming input they use (mouse and keyboard or controller), gaming experience, and any self-reported symptoms of musculoskeletal issues from prolonged gaming if any.
3. Potential participants will be contacted within 48 hours of completing the demographic survey informing them of whether or not they are eligible.
4. Eligible participants will complete informed consent via Zoom after 3 days of being informed of eligibility for the study by the student researcher 1 week prior to beginning the study. Potential participants will have 48 hours to make a decision on whether or not they would like to participate in the study.
5. Week Zero of the study will commence and baseline assessments will be performed in person at either Black Fire Innovation or the Tonopah Lounge based on participate convenience, using REBA to assess ergonomic risks and Kovaaks to assess current gaming performance. A questionnaire exploring their current knowledge via Qualtrics in ergonomics will also be provided during this first visit. Participants will be given a scheduled time to show up for this part of data collection.
6. During week one, the student researcher will deliver the supplemental educational component and the ergonomic protocol in person at the Tonapah Lounge. The educational module and ergonomic protocol will be attached. This session will approximately take about 45 minutes to an hour to deliver all information. All information will be found on a website created by the student researcher as a hub for all information taught and implemented during this visit. Handouts of the protocol will also be provided.
7. During week three, the student researcher will conduct an in-person follow-up at the Tonapah Lounge or Black Fire Innovation depending on participant convenience assessing any changes in ergonomic risk and performance using REBA and Kovaaks which will approximately take about 60-90 minutes. Participants will be given a scheduled time to show up for this part of data collection.
8. A second in-person follow-up will be conducted during week six using REBA and Kovaaks, and the focus group will be conducted at this time to explore their progress in the implementation of the protocol after gathering all objective data. This focus group will comprise of 5-7 volunteer participants who will be provided with an incentive of an additional $10 gift card to Steam, a gaming platform. This focus group will be conducted in a secure room at the Tonapah Lounge, separate from the shared space area. An audio recording of the session will be done for the duration of the session for the purpose of transcription. Participants will be assigned unique identifiers to uphold privacy and confidentiality. An audio recording of the session will be done on a password-protected device.
9. A post-survey will also be distributed to all participants via Qualtrics at Week 6. This will take a total of 2-3 hours for the visit.
10. A long-term follow-up will be conducted at Week 12. Participants will receive a questionnaire created on Qualtrics via email to explore adherence to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Primarily participates in PC games(s) using mouse and keyboard for at least a year
* Plays at least 10 hours a week
* Must be affiliated with an established Esports team or organization
* Must have transportation

Exclusion Criteria:

* Individuals currently receiving treatment for self-reported pain related to prolonged gaming
* Those with a history of surgical procedures in the upper extremities
* Individuals with cognitive impairments
* Individuals with a history of a neck, shoulder, wrist, and/or back injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Rapid Entire Body Assessment (REBA) | At intervals throughout the 6 week cycle.
  The REBA is a standardized ergonomic assessment tool used to evaluate the risk of musculoskeletal strain associated with specific body postures and tasks. In this study, the REBA is used to analyze the participants' gaming postures, focusing on key areas such as the neck, back, shoulders, arms, and wrists. Scores are generated based on observed postures and movements, with higher scores indicating greater ergonomic risk. This outcome measure helps identify and quantify changes in participants' ergonomic risk levels before, during, and after the intervention.
Kovaaks | At intervals throughout the 6 week cycle.
  Kovaaks is a gaming performance training and evaluation software designed for esports athletes. It provides customizable scenarios to assess and improve critical gaming skills, such as aim, accuracy, and reaction time. In this study, Kovaaks is used as an objective measure to track changes in participants' gaming performance over the six-week protocol. Metrics such as actions per minute (APM), accuracy percentages, and reaction times are recorded to evaluate the impact of the ergonomic intervention on performance outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Breach of informed consent.

REFERENCES:
- See also: Information hub including educational component of the study and the protocol. — https://rivera2183.wixsite.com/level-up-gaming